CLINICAL TRIAL: NCT01225055
Title: Effect of Teriparatide, Vibration and the Combination on Bone Mass and Bone Architecture in Chronic Spinal Cord Injury
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Thomas J. Schnitzer (Other)
Collaborators: Edward Hines Jr. VA Hospital (U.S. Federal Agency); University of Illinois at Chicago (Other); Congressionally Directed Medical Research Program (Unknown)
Responsible Party: Sponsor-Investigator, Thomas J. Schnitzer, professor, Northwestern University
Organization: Northwestern University (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: STU00033380; CDMRP-SC090010 (Other Grant/Funding Number: Department of Defense)
Record Dates: First submitted 2010-10-19; First posted 2010-10-20 (Estimated); Results first posted 2017-06-22 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-11

CONDITIONS: Spinal Cord Injury; Bone Loss; Osteoporosis
MeSH Terms: conditions — Spinal Cord Injuries; Bone Diseases, Metabolic; Osteoporosis | interventions — Teriparatide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Teriparatide (Experimental): Teriparatide alone with sham vibration
  Interventions: Drug: Teriparatide
- Vibration (Experimental): Vibration alone with placebo-teriparatide
  Interventions: Device: vibration
- Teriparatide and vibration (Experimental): Teriparatide with vibration applied in conjuction
  Interventions: Drug: Teriparatide; Device: vibration

INTERVENTIONS:
Drug: Teriparatide — 20 ug daily over 12 months
  Other Names: Forteo
  Arms: Teriparatide; Teriparatide and vibration
Device: vibration — 10 min/day for 12 months
  Arms: Teriparatide and vibration; Vibration

SUMMARY:
Spinal cord injury (SCI) results in marked acute loss of bone. This study evaluates the effect of teriparatide (PTH) and the use of vibration as a form of mechanical stimulation on bone mass.

DETAILED DESCRIPTION:
The aim of this study is to evaluate PTH with vibration in a group of individuals with chronic SCI and loss of bone mass in their lower extremities. A convenience sample of 60 subjects with SCI will be enrolled into a 12 month study assessing the effects of PTH (20 ug/day) and vibration (10 min/day) individually or in combination on BMD and bone markers. Subjects will be evaluated at 3, 6, 9, and 12 months after initiating treatment with measurement of bone density as well as bone markers of formation and resorption.

ELIGIBILITY:
Inclusion Criteria:

Age >21 years (must have closed epiphyses; PTH contraindicated if epiphyses open)

* Both males and females
* SCI with inability to ambulate independently
* Capable of positioning to have DXA performed
* Low bone mass at the total hip by DEXA (Z score < 1.5; T score < 2.5 or T score <-2.0 plus preexisting fragility fracture)
* Capable of reading and understanding informed consent document
* Able to self-administer teriparatide or have someone in the family who can do so
* No known endocrinopathies
* Normal TSH levels
* Normal 25-OH vitamin D levels (> 30ng/ml)
* Normal calcium levels
* Normal renal function (creatinine <2.0mg/dl)
* Able to return for all follow-up visits

Exclusion Criteria:

Surgical or other intervention resulting in metal or anatomy precluding obtaining DXA measurements (e.g., cardiac pacemakers, ferromagnetic implants or brain aneurysm clips).

* Had had an allergic reaction to Teriparatide (FORTEO) or one of its ingredients.
* Have Paget's disease of the bone
* Have unexplained high levels of f alkaline phosphatase in blood
* Any active Gastrointestinal condition that results in malabsorption
* History of presence of alcoholism or drug abuse within the 2 years prior to study screening
* Other medical conditions that in the opinion of the investigator would preclude the subject from completing the study
* History of malignancy. Patients having had basal cell carcinomas successfully removed will be allowed to enroll in the protocol.
* History of radiation therapy
* Unable to self-administer PTH or have it administered
* Elevated liver function tests >2x normal
* Currently being prescribed anti-convulsants
* Currently being prescribed glucocorticoids, other than inhaled glucocorticoids
* Currently being prescribed any bone-active agents, including any bisphosphonate, raloxifene, hormone therapy (estrogen and estrogen/progestin), calcitonin or strontium-containing compounds. Bisphosphonate use will be allowed up the time of initiation of study medication but not during the dosing with study medication.
* Previous history of PTH use
* Pregnant, planning to become pregnant, or lactating

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2010-10; Primary Completion 2015-08 (Actual); Study Completion 2016-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas J Schnizter, MD, PhD, Principal Investigator — Northwestern University
Locations (2):
- United States (2):
  - Northwestern University Feinberg School of Medicine, Chicago, Illinois
  - Edward Hines, Jr, VA Hospital, Maywood, Illinois

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Haider IT, Lobos SM, Simonian N, Schnitzer TJ, Edwards WB. Bone fragility after spinal cord injury: reductions in stiffness and bone mineral at the distal femur and proximal tibia as a function of time. Osteoporos Int. 2018 Dec;29(12):2703-2715. doi: 10.1007/s00198-018-4733-0. Epub 2018 Oct 17. PMID 30334093

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: One subject withdrew prior to receiving therapy from the "Teriparatide and Vibration" group. After consenting the subject did not participate in the study.. This accounts for the 61 in Participant Flow but 60 that were enrolled and started treatment according to their assigned group.
Period: Overall Study
Arm/Group | Teriparatide | Vibration | Teriparatide and Vibration
Started | 20 | 20 | 21
Completed | 20 | 18 | 18
Not Completed | 0 | 2 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Teriparatide | Vibration | Teriparatide and Vibration | Total
Number analyzed (Participants) | 20 | 20 | 21 | 61
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 16 | 18 | 19 | 53
  >=65 years | 4 | 2 | 2 | 8
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.6 (16.3) | 40.9 (16.4) | 46.6 (15.4) | 45.4 (16.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 6 | 5 | 14
  Male | 17 | 14 | 16 | 47
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 4 | 6 | 16
  Not Hispanic or Latino | 14 | 16 | 15 | 45
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 2 | 0 | 2
  Black or African American | 9 | 10 | 14 | 33
  White | 11 | 7 | 7 | 25
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 20 | 20 | 21 | 60

OUTCOME MEASURES:

1. Primary Outcome: Bone Mineral Density BMD of the Total Hip as Assessed by DXA.
Description: The mean change in BMD of the total hip after 12 month of treatment
Time Frame: Baseline to 12 Months
Population: One subject withdrew prior to receiving therapy. The samples from the Hines location (n=11) were also not included. Two additional subjects were not analyzed due to metal artifacts or heterotopic ossification that interfered with analysis. This accounts for the 14 subjects that were not analyzed.
Measure: Mean (Standard Deviation); unit: g/cm^2
Arm/Group | Teriparatide | Vibration | Teriparatide and Vibration
Number analyzed (Participants) | 15 | 17 | 15
g/cm^2
  0 months | 0.66 (0.03) | 0.63 (0.03) | 0.64 (0.03)
  3 months | 0.65 (0.03) | 0.63 (0.03) | 0.65 (0.03)
  6 months | 0.67 (0.03) | 0.63 (0.03) | 0.65 (0.03)
  12 months | 0.66 (0.03) | 0.64 (0.03) | 0.65 (0.03)
Statistical Analysis 1: Comparison: Teriparatide vs Vibration vs Teriparatide and Vibration; Test type: Superiority; p = 0.84, ANOVA — calculated p-value indicating the effect of different treatment groups; Repeated measures ANOVA
Statistical Analysis 2: Comparison: Teriparatide vs Vibration vs Teriparatide and Vibration; Test type: Superiority; p = 0.64, ANOVA — calculated p-value indicating the effect of different time points; Repeated measures ANOVA
Statistical Analysis 3: Comparison: Teriparatide vs Vibration vs Teriparatide and Vibration; Test type: Superiority; p = 0.26, ANOVA — calculated p-value indicating the effect of different treatment groups and time points; Repeated measures ANOVA

2. Secondary Outcome: Bone Mineral Density (BMD) by DXA at the Lumbar Spine.
Description: The mean change in BMD at the lumbar spine from baseline after 12 month of treatment
Time Frame: Baseline to 12 Months
Population: One subject withdrew prior to receiving therapy. The samples from the Hines location (n=11) were also not included. Five additional subjects were not analyzed due to metal artifacts that interfered with analysis. This accounts for the 17 subjects that were not analyzed.
Measure: Mean (Standard Deviation); unit: g/cm^2
Arm/Group | Teriparatide | Vibration | Teriparatide and Vibration
Number analyzed (Participants) | 16 | 14 | 14
g/cm^2
  0 months | 1.04 (0.04) | 1.00 (0.04) | 1.02 (0.04)
  3 months | 1.05 (0.04) | 1.01 (0.04) | 1.04 (0.04)
  6 months | 1.07 (0.04) | 1.02 (0.04) | 1.05 (0.04)
  12 months | 1.09 (0.04) | 1.02 (0.04) | 1.07 (0.04)
Statistical Analysis 1: Comparison: Teriparatide vs Vibration vs Teriparatide and Vibration; Test type: Superiority; p = 0.64, ANOVA — calculated p-value indicating the effect of different treatment groups; Repeated measures ANOVA
Statistical Analysis 2: Comparison: Teriparatide vs Vibration vs Teriparatide and Vibration; Test type: Superiority; p = 0.00, ANOVA — calculated p-value indicating the effect of different time points; Repeated measures ANOVA
Statistical Analysis 3: Comparison: Teriparatide vs Vibration vs Teriparatide and Vibration; Test type: Superiority; p = 0.09, ANOVA — calculated p-value indicating the effect of different treatment groups and time points; Repeated measures ANOVA

3. Secondary Outcome: Bone Mineral Density (BMD) by DXA at Femoral Neck
Description: The mean change in BMD of the femoral neck after 12 month of treatment
Time Frame: Baseline to 12 Months
Population: One subject withdrew prior to receiving therapy. The samples from the Hines location (n=11) were also not included. One additional subjects was not analyzed due to metal artifacts or heterotopic ossification that interfered with analysis. This accounts for the 13 subjects that were not analyzed.
Measure: Mean (Standard Deviation); unit: g/cm^2
Arm/Group | Teriparatide | Vibration | Teriparatide and Vibration
Number analyzed (Participants) | 15 | 17 | 16
g/cm^2
  0 months | 0.66 (0.03) | 0.63 (0.03) | 0.62 (0.03)
  3 months | 0.66 (0.04) | 0.64 (0.04) | 0.63 (0.04)
  6 months | 0.67 (0.04) | 0.62 (0.03) | 0.63 (0.04)
  12 months | 0.66 (0.03) | 0.63 (0.03) | 0.63 (0.03)
Statistical Analysis 1: Comparison: Teriparatide vs Vibration vs Teriparatide and Vibration; Test type: Superiority; p = 0.72, ANOVA — calculated p-value indicating the effect of different treatment groups; Repeated measures ANOVA
Statistical Analysis 2: Comparison: Teriparatide vs Vibration vs Teriparatide and Vibration; Test type: Superiority; p = 0.58, ANOVA — calculated p-value indicating the effect of different time points; Repeated measures ANOVA
Statistical Analysis 3: Comparison: Teriparatide vs Vibration vs Teriparatide and Vibration; Test type: Superiority; p = 0.44, ANOVA — calculated p-value indicating the effect of different treatment groups and time points; Repeated measures ANOVA

4. Secondary Outcome: C-terminal Telopeptide
Description: The mean change in C-terminal telopeptide from baseline after 12 month of treatment
Time Frame: Baseline to 12 Months
Population: One subject withdrew prior to receiving therapy from the Teriparatide and Vibration group. One sample was lost due to laboratory error. The samples from the Hines location (n=11) were also not included in this analysis. This accounts for the 13 subjects that were not analyzed.
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Teriparatide | Vibration | Teriparatide and Vibration
Number analyzed (Participants) | 15 | 17 | 16
ng/ml
  0 months | 0.38 (0.07) | 0.31 (0.06) | 0.38 (0.06)
  3 months | 0.72 (0.11) | 0.25 (0.10) | 0.43 (0.11)
  6 months | 0.74 (0.11) | 0.25 (0.11) | 0.44 (0.11)
  12 months | 0.59 (0.11) | 0.29 (0.11) | 0.45 (0.11)
Statistical Analysis 1: Comparison: Teriparatide vs Vibration vs Teriparatide and Vibration; Test type: Superiority; p = 0.02, ANOVA — calculated p-value indicating the effect of different treatment groups; Repeated measures ANOVA
Statistical Analysis 2: Comparison: Teriparatide vs Vibration vs Teriparatide and Vibration; Test type: Superiority; p = 0.10, ANOVA — calculated p-value indicating the effect of different time points; Repeated measures ANOVA
Statistical Analysis 3: Comparison: Teriparatide vs Vibration vs Teriparatide and Vibration; Test type: Superiority; p = 0.04, ANOVA — calculated p-value indicating the effect of different treatment groups and time points; Repeated measures ANOVA

5. Secondary Outcome: Bone-specific Alkaline Phosphatase
Description: The mean change in Bone-specific alkaline phosphatase from baseline after 12 month of therapy
Time Frame: Baseline to 12 Months
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Teriparatide | Vibration | Teriparatide and Vibration
Number analyzed (Participants) | 15 | 17 | 16
ng/ml
  0 months | 15.3 (1.63) | 13.9 (1.53) | 12.4 (1.58)
  3 months | 18.4 (1.81) | 11.6 (1.70) | 12.8 (1.75)
  6 months | 20.3 (2.64) | 11.3 (2.48) | 16.2 (2.56)
  12 months | 20.4 (1.58) | 11.8 (1.48) | 14.0 (1.53)
Statistical Analysis 1: Comparison: Teriparatide vs Vibration vs Teriparatide and Vibration; Test type: Superiority; p = 0.01, ANOVA — calculated p-value indicating the effect of different treatment groups; Repeated measures ANOVA
Statistical Analysis 2: Comparison: Teriparatide vs Vibration vs Teriparatide and Vibration; Test type: Superiority; p = 0.34, ANOVA — calculated p-value indicating the effect of different time points; Repeated measures ANOVA
Statistical Analysis 3: Comparison: Teriparatide vs Vibration vs Teriparatide and Vibration; Test type: Superiority; p = 0.20, ANOVA — calculated p-value indicating the effect of different treatment groups and time points; Repeated measures ANOVA

6. Secondary Outcome: Amino-terminal Propeptide of Type 1 Collagen
Description: The mean change in Amino-terminal of type 1 collagen from baseline after 12 months of treatment
Time Frame: Baseline to 12 Months
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Teriparatide | Vibration | Teriparatide and Vibration
Number analyzed (Participants) | 15 | 17 | 16
ng/ml
  0 months | 67.1 (8.90) | 64.7 (8.36) | 67.9 (8.61)
  3 months | 128 (12.9) | 51.8 (12.1) | 90.1 (12.5)
  6 months | 163 (30.4) | 54.5 (28.6) | 125 (29.4)
  12 months | 124 (13.5) | 49.8 (12.7) | 77.0 (13.0)
Statistical Analysis 1: Comparison: Teriparatide vs Vibration vs Teriparatide and Vibration; Test type: Superiority; p = 0.00, ANOVA — calculated p-value indicating the effect of different treatment groups; Repeated measures ANOVA
Statistical Analysis 2: Comparison: Teriparatide vs Vibration vs Teriparatide and Vibration; Test type: Superiority; p = 0.01, ANOVA — calculated p-value indicating the effect of different time points; Repeated measures ANOVA
Statistical Analysis 3: Comparison: Teriparatide vs Vibration vs Teriparatide and Vibration; Test type: Superiority; p = 0.04, ANOVA — calculated p-value indicating the effect of different treatment groups and time points; Repeated measures ANOVA

ADVERSE EVENTS:
Time Frame: Baseline to 12 months
Description: One subject withdrew prior to receiving therapy from the "Teriparatide and Vibration" group. The adverse events for this individual were not reported. This explains why for the "Teriparatide and Vibration" n = 20 rather than n = 21.
Arm/Group | Teriparatide | Vibration | Teriparatide and Vibration
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/20 | 0/20
Serious Adverse Events (participants affected / at risk) | 7/20 | 1/20 | 8/20
Other Adverse Events (participants affected / at risk) | 16/20 | 16/20 | 16/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Teriparatide (N=20) | Vibration (N=20) | Teriparatide and Vibration (N=20)
Cardiovascular Event (Cardiac disorders) | 1 (3) | 0 (0) | 0 (0)
Injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 2 (2)
Lower extremity fracture (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0)
Pneumonia and respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (4)
Soft tissue infection (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 2 (2)
Urinary tract infection (Renal and urinary disorders) | 4 (5) | 1 (1) | 2 (8)
OTHER ADVERSE EVENTS (reported when occurring in more than 5.0% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Teriparatide (N=20) | Vibration (N=20) | Teriparatide and Vibration (N=20)
Acid Reflux (Gastrointestinal disorders) | 4 (4) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 (6) | 1 (1) | 4 (6)
Bleeding, bruising or irritation at injection site (Skin and subcutaneous tissue disorders) | 3 (3) | 3 (3) | 6 (6)
Burns (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 2 (2)
Chest Pain (Cardiac disorders) | 0 (0) | 1 (1) | 1 (2)
Constipation (Gastrointestinal disorders) | 4 (4) | 5 (5) | 2 (2)
Dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 5 (5) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 2 (2) | 1 (1) | 1 (1)
Dizziness (Nervous system disorders) | 2 (2) | 3 (3) | 7 (8)
Flu like symptoms (Infections and infestations) | 5 (6) | 2 (2) | 2 (4)
Headache (Nervous system disorders) | 2 (2) | 3 (4) | 4 (4)
Increased Nerve Pain (Nervous system disorders) | 2 (2) | 0 (0) | 2 (3)
Increased spasticity (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2)
Indigestion (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2)
Injury (Injury, poisoning and procedural complications) | 2 (2) | 3 (5) | 4 (4)
Lower extremity fractures (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2) | 1 (1)
Lower extremity pain (Musculoskeletal and connective tissue disorders) | 4 (5) | 0 (0) | 1 (2)
Nausea/Vomitting (Gastrointestinal disorders) | 4 (4) | 3 (3) | 4 (5)
Parageusia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2)
Parathesias (Nervous system disorders) | 2 (2) | 0 (0) | 2 (2)
Pressure sore (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 3 (7)
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2)
Upper respiratory infection (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 5 (6) | 5 (6)
Urinary tract infection (Renal and urinary disorders) | 9 (11) | 3 (4) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No